CLINICAL TRIAL: NCT07144787
Title: Patient Satisfaction and Oral Health Related Quality of Life for Four Implant Retained Mandibular Overdenture VERSUS Fixed-detachable Prosthesis. Crossover Clinical Study
Brief Title: Four Implant Retained Mandibular Overdenture VERSUS Fixed-detachable Prosthesis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A02010024RP
Record Dates: First submitted 2025-08-25; First posted 2025-08-28 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-08

CONDITIONS: Oral Health Impact Profile Short Version 14 (OHIP 14)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- implant retained complete Overdenture (Active Comparator): implant retained complete Overdenture
  Interventions: Other: implant retained complete Overdenture
- Fixed-detachable prosthesis. (Active Comparator): Fixed-detachable prosthesis.
  Interventions: Other: Fixed-detachable prosthesis

INTERVENTIONS:
Other: implant retained complete Overdenture — four implant retained complete Overdenture versus Fixed-detachable prosthesis
  Arms: implant retained complete Overdenture
Other: Fixed-detachable prosthesis — four implant retained complete Overdenture versus Fixed-detachable prosthesis.
  Arms: Fixed-detachable prosthesis.

SUMMARY:
ABSTRACT Statement of the problem: completely edentulous patient can be treated by four implants for implant retained overdenture or fixed detachable prosthesis.

Purpose: the purpose of this clinical study is to evaluate patient satisfaction and oral health impact profile (OHIP-14) for four implant retained complete Overdenture versus Fixed-detachable prosthesis.

Material and methods: This clinical cross-over study included 10 completely edentulous patients with maxillary single denture and four parallel implants were placed intraforminal. Every patient received two mandibular implants at the 1st premolar region and two mandibular implants in lateral incisor region. Ten completely edentulous patients received implant retained overdenture for six months (Group I), then fixed detachable prostheses on four implants for the following six months (Group II). For both designs, patient satisfaction using visual analogue scale (VAS) and oral health impact profile (OHIP-14) will be recorded for both prostheses. SPSS program will be used for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:
* This research will be done on patients who were previously received 2 mesially placed implants in the 1st premolar region with only two remaining mandibular canines with opposing maxillary single denture

Exclusion Criteria:

* uncontrolled diabetic patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-01-12 (Actual)

PRIMARY OUTCOMES:
patients indicated satisfaction with their prosthesis using a visual analog scale (VAS) | 6 months
  participants will be asked to score their answer according to the amount of satisfaction on a 100 mm line (Score 0 = no satisfaction at all and score 100 = complete satisfaction).

SECONDARY OUTCOMES:
oral health impact profile (OHIP-14) was recorded for both prostheses. | 6 months
  Regarding the oral health-related quality of life (OHRQoL), oral health impact profile (OHIP-14), the questions covered seven domains: functional limitation, physical pain, physical disability, psychologic discomfort, psychologic disability, social disability, and handicap. Also, these questions will be translated into Arabic by linguistic professionals who act in collaboration with the authors to prepare the final version. The translation will be made using a forward-backward approach. The answers of the questionnaire include score 1 = never, score 2 = hardly ever, score 3 = occasionally, score 4 = fairly often, and score 5 = very often.

CONTACTS AND LOCATIONS:
Locations (1):
- Basmsa, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided